CLINICAL TRIAL: NCT05878197
Title: Effect of Semi-occluded Vocal Tract Therapy on the Phonation of Children With Vocal Fold Nodules.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B670201936069 (BC-04563)
Record Dates: First submitted 2023-04-18; First posted 2023-05-26 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Voice Disorders in Children; Vocal Nodules in Children; Hoarseness; Dysphonia
Keywords: semi-occluded vocal tract therapy; straw phonation; resonant voice therapy; vocal hygiene
MeSH Terms: conditions — Hoarseness; Dysphonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 - Straw Phonation (Experimental): Short-term intensive voice therapy program of one week (3 hours a day for 4 consecutive days): straw phonation and vocal hygiene recommendations
  Interventions: Behavioral: Straw phonation
- Experimental group 2 - Resonant Voice Therapy (Experimental): Short-term intensive voice therapy program of one week (3 hours a day for 4 consecutive days): resonant voice therapy and vocal hygiene recommendations
  Interventions: Behavioral: Resonant voice therapy
- Control group (Sham Comparator): Short-term intensive voice therapy program of one week (3 hours a day for 4 consecutive days): vocal hygiene recommendations
  Interventions: Behavioral: Vocal Hygiene

INTERVENTIONS:
Behavioral: Straw phonation — The two experimental groups will receive either straw phonation therapy or resonant voice therapy. The hierarchical structure of the therapy sessions will be equal for the three programs. In each session, vocal rest pauses will be foreseen by playing games, performing drawing assignments, etc. This will make the therapy more pleasant and less intensive. All voice therapy programs will be guided by the same experienced voice therapist.
  Content:
  Day 1: counseling (anatomy and physiology of the voice and vocal fold nodules), vocal hygiene recommendations (water intake, avoiding vocal misuse and abuse) Day 2: breathing exercises, vocal hygiene recommendations, straw phonation on vowel and syllable level, pitch variations Day 3: breathing exercises, vocal hygiene recommendations, straw phonation on word and sentence level, pitch variations Day 4: straw phonation in spontaneous speech, combination exercises
  Arms: Experimental group 1 - Straw Phonation
Behavioral: Resonant voice therapy — The two experimental groups will receive either straw phonation therapy or resonant voice therapy. The hierarchical structure of the therapy sessions will be equal for the three programs. In each session, vocal rest pauses will be foreseen by playing games, performing drawing assignments, etc. This will make the therapy more pleasant and less intensive. All voice therapy programs will be guided by the same experienced voice therapist.
  Content:
  Day 1: counseling (anatomy and physiology of the voice and vocal fold nodules), vocal hygiene recommendations (water intake, avoiding vocal misuse and abuse) Day 2: breathing exercises, vocal hygiene recommendations, resonant voice therapy on vowel and syllable level, pitch variations Day 3: breathing exercises, vocal hygiene recommendations, resonant voice therapy on word and sentence level, pitch variations Day 4: resonant voice therapy in spontaneous speech, combination exercises
  Arms: Experimental group 2 - Resonant Voice Therapy
Behavioral: Vocal Hygiene — Participants of the control group will receive a sham treatment, including the exact same games, drawing assignments, etc. as in the experimental groups. However, no SOVT or other active vocal techniques will be practiced. Vocal hygiene guidelines (e.g. avoid screaming, imitating voices, sufficient hydration etc.) will be kept equally in the four groups. All voice therapy programs will be guided by the same experienced voice therapist.
  Content:
  Day 1: counseling (anatomy and physiology of the voice and vocal fold nodules), vocal hygiene recommendations (water intake, avoiding vocal misuse and abuse) Day 2: breathing exercises, vocal hygiene recommendations Day 3: breathing exercises, vocal hygiene recommendations Day 4: combination exercises
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to determine and compare the effects of different voice therapy programs in children with vocal fold nodules. Vocal fold nodules are non-cancerous growths on the vocal folds which cause hoarseness. The main questions this trial aims to answer are:

* What are the short-term effects of the new voice therapy program 'straw phonation' and a more traditional 'resonant voice therapy' program on (a) the vocal quality, (b) the size of the growths on the vocal folds, and (c) the overall functioning in children with vocal fold nodules? During straw phonation exercises, you make sound through a drinking straw. During resonant voice therapy exercises or 'humming', you make an 'm' sound as you breathe out.
* What are the long-term effects of these voice therapy programs?

Participants will receive a short-term intensive voice therapy program of four days. The researchers will compare the straw phonation group, resonant voice therapy group and control group to see if voice therapy works well in treating children with vocal fold nodules.

The researchers hypothesize that straw phonation will have better results than resonant voice therapy. Straw phonation exercises are easier for children because they use an external tool (the straw) and less self-correction is needed.

DETAILED DESCRIPTION:
Background:

The main goal of voice therapy in children with vocal fold nodules is to improve their communication, vocal quality and wellbeing. However, in this population, efficacy or effectiveness studies of voice therapy are extremely limited and show methodological shortcomings. There is an urgent need to understand the impact of different semi-occluded vocal tract (SOVT) techniques on the multidimensional facets of voice, as these SOVT exercises are frequently used in clinical practice. The common feature of these exercises is a reduction in the cross-sectional area of the vocal tract while voicing. Results of this project will have an impact on evidence-based voice therapy in children and consequently on reimbursement agreements of the health care system in the future. This fundamental research regarding the impact of SOVT techniques on the voice can also lead to the development and improvement of SOVT techniques.

Purposes:

* The first purpose of this project is to determine and compare the short-term effect of a "non-intuitive" SOVT therapy program (straw phonation) with a more traditional "intuitive" resonant voice therapy program of one week on (a) the vocal quality, (b) the laryngeal anatomy and function, and (c) the psychosocial wellbeing in children (aged between 6 and 12 years) with vocal fold nodules using a randomized sham-controlled trial.
* The second purpose of this project is to determine and compare the long-term effect of these voice therapy programs on (a) the vocal quality, (b) the laryngeal anatomy and function, and (c) the psychosocial wellbeing of the children.

Hypotheses:

Giving the promising physics of an SOVT, a positive short-term effect of straw phonation and resonant voice therapy is hypothesized. However, the non-intuitive technique straw phonation is expected to be in favor for a pediatric population. For these exercises, semi-occlusions are created by an external tool and instructions, feedback, and self-corrections can be reduced to a minimum. These factors might lead to faster results, which might in turn reduce feelings of frustration and demotivation by the children.

Study design:

A longitudinal randomized sham-controlled trial will be used. Patients will be randomly assigned to one of the 2 treatment groups "straw phonation", "resonant voice therapy", or the control group receiving a "sham treatment".

Innovativity:

This research will be innovative because of (a) the topic and study population (SOVT in children between 6 and 12 years) which is an underexposed domain in literature; (b) the methods investigating multidimensional facets of voice (c) the randomized sham-controlled study design using a large study group, a control group receiving sham treatment, random allocation of participants and blinded assessors and (d) the combination of short-term and long-term outcome.

Participants:

Inclusion criteria and exclusion criteria are described further in the application.

Voice assessment:

A standardized and multidimensional voice assessment including both objective and subjective vocal outcomes will be performed to evaluate the participants' voice pre and post-therapy, and at 3 months and 6 months follow-up. The multidimensional voice assessment will consist of the following outcomes: (a) vocal quality, (b) laryngeal anatomy and function, and c) psychosocial wellbeing. Assessments (a) and (c) will be performed in a sound-treated room at Ghent University Hospital by speech-language pathologists experienced in voice diagnostics. Assessments (b) will be performed by experienced otorhinolaryngologist. All assessors will be blinded to group allocation and study evolution. A detailed overview of the outcome characteristics is described further in the application.

Voice therapy:

The content of the different therapy arms / interventions is described further in the application.

Statistical analysis:

Linear mixed model analyses (LMM) will be used to determine whether there is a difference in evolution between the groups over time. Post-hoc pairwise comparisons with Bonferroni corrections will uncover specific within and between group differences. Intraclass correlation coefficients models and Cohen's κ will be used to determine inter- ant intrarater reliability.

ELIGIBILITY:
Inclusion Criteria:

* children aged between 6 and 12 years (primary school)
* diagnosed with vocal fold nodules by an otorhinolaryngologist and speech-language pathologist experienced in voice diagnostics.

Exclusion Criteria:

* nasal or ear diseases
* neurological disorders

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristiane Van Lierde, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartnick C, Ballif C, De Guzman V, Sataloff R, Campisi P, Kerschner J, Shembel A, Reda D, Shi H, Sheryka Zacny E, Bunting G. Indirect vs Direct Voice Therapy for Children With Vocal Nodules: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Feb 1;144(2):156-163. doi: 10.1001/jamaoto.2017.2618. PMID 29270612
- [Background] Kapsner-Smith MR, Hunter EJ, Kirkham K, Cox K, Titze IR. A Randomized Controlled Trial of Two Semi-Occluded Vocal Tract Voice Therapy Protocols. J Speech Lang Hear Res. 2015 Jun;58(3):535-49. doi: 10.1044/2015_JSLHR-S-13-0231. PMID 25675335
- [Background] Carding PN, Roulstone S, Northstone K; ALSPAC Study Team. The prevalence of childhood dysphonia: a cross-sectional study. J Voice. 2006 Dec;20(4):623-30. doi: 10.1016/j.jvoice.2005.07.004. Epub 2005 Dec 19. PMID 16360302
- [Background] Meerschman I, Van Lierde K, Van Puyvelde C, Bostyn A, Claeys S, D'haeseleer E. Massed versus spaced practice in vocology: effect of a short-term intensive voice training versus a longer-term traditional voice training. Int J Lang Commun Disord. 2018 Mar;53(2):393-404. doi: 10.1111/1460-6984.12358. Epub 2017 Dec 5. PMID 29205707

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group 1 - Straw Phonation: Short-term intensive voice therapy program of one week (3 hours a day for 4 consecutive days): straw phonation and vocal hygiene recommendations
  Straw phonation: The two experimental groups received either straw phonation therapy or resonant voice therapy. The hierarchical structure of the therapy sessions was equal for the three programs. In each session, vocal rest pauses were foreseen by playing games, performing drawing assignments, etc. This made the therapy more pleasant and less intensive. All voice therapy programs were guided by the same experienced voice therapist.
  Content:
  Day 1: counseling (anatomy and physiology of the voice and vocal fold nodules), vocal hygiene recommendations (water intake, avoiding vocal misuse and abuse) Day 2: breathing exercises, vocal hygiene recommendations, straw phonation on vowel and syllable level, pitch variations Day 3: breathing exercises, vocal hygiene recommendations, straw phonation on word and sentence level, pitch variations Day 4: straw phonation in spontaneous speech, combination exercises
- Experimental Group 2 - Resonant Voice Therapy: Short-term intensive voice therapy program of one week (3 hours a day for 4 consecutive days): resonant voice therapy and vocal hygiene recommendations
  Resonant voice therapy: The two experimental groups received either straw phonation therapy or resonant voice therapy. The hierarchical structure of the therapy sessions was equal for the three programs. In each session, vocal rest pauses were foreseen by playing games, performing drawing assignments, etc. This made the therapy more pleasant and less intensive. All voice therapy programs were guided by the same experienced voice therapist.
  Content:
  Day 1: counseling (anatomy and physiology of the voice and vocal fold nodules), vocal hygiene recommendations (water intake, avoiding vocal misuse and abuse) Day 2: breathing exercises, vocal hygiene recommendations, resonant voice therapy on vowel and syllable level, pitch variations Day 3: breathing exercises, vocal hygiene recommendations, resonant voice therapy on word and sentence level, pitch variations Day 4: resonant voice therapy in spontaneous speech, combination exercises
- Control Group: Short-term intensive voice therapy program of one week (3 hours a day for 4 consecutive days): vocal hygiene recommendations
  Vocal Hygiene: Participants of the control group received a sham treatment, including the exact same games, drawing assignments, etc. as in the experimental groups. However, no SOVT or other active vocal techniques were practiced. Vocal hygiene guidelines (e.g. avoid screaming, imitating voices, sufficient hydration etc.) were kept equally in the three groups. All voice therapy programs were guided by the same experienced voice therapist.
  Content:
  Day 1: counseling (anatomy and physiology of the voice and vocal fold nodules), vocal hygiene recommendations (water intake, avoiding vocal misuse and abuse) Day 2: breathing exercises, vocal hygiene recommendations Day 3: breathing exercises, vocal hygiene recommendations Day 4: combination exercises
Period: Overall Study
Arm/Group | Experimental Group 1 - Straw Phonation | Experimental Group 2 - Resonant Voice Therapy | Control Group
Started | 11 | 11 | 8
Completed | 11 | 11 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group 1 - Straw Phonation | Experimental Group 2 - Resonant Voice Therapy | Control Group | Total
Number analyzed (Participants) | 11 | 11 | 8 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 11 | 8 | 30
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.55 (2.2) | 8.79 (1.5) | 9.21 (1.9) | 8.81 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 3 | 14
  Male | 6 | 5 | 5 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 11 | 11 | 8 | 30
Dysphonia Severity Index [Mean (Standard Deviation); unit: units on a scale] — The Dysphonia Severity Index is calculated using the following formula: 0.13 × MFT + 0.0053 × fhigh - 0.26 × Ilow - 1.18 × jitter + 12.4. The index value obtained usually ranges between -5 and +5. A lower index value indicates poorer vocal quality or, more generally, poorer vocal functioning (Awan & Ensslen, 2010). The threshold score that distinguishes a normophonic from a dysphonic voice is 1.6 (Raes et al., 2002).
  units on a scale | -3.0 (3.3) | -2.6 (2.8) | -2.5 (3.2) | -2.7 (3.0)
Acoustic Voice Quality Index [Mean (Standard Deviation); unit: units on a scale] — The Acoustic Voice Quality Index (AVQI) is an objective, multiparameter approach to quantify dysphonia severity on the basis of a sustained vowel [a:] and continuous speech (Maryn, Corthals, et al., 2010). The formula of the AVQI is 2.571 (3.295 - 0.111 CPPs - 0.073 HNR - 0.213 SL + 2.789 SLdB - 0.032 slope + 0.077 tilt). The index ranges from 0 to 10 and a higher index indicates poorer vocal quality. The threshold score that distinguishes a normophonic voice from a dysphonic voice in Dutch is 2.95 (Maryn, Corthals, et al., 2010).
  units on a scale | 4.16 (1.5) | 4.50 (1.4) | 4.37 (1.2) | 4.34 (1.4)
Pediatric Voice Handicap Index [Mean (Standard Deviation); unit: units on a scale] — A parent completed the Dutch version of the pVHI, which is a parent-proxy tool to gain insight into the physical, functional and emotional impact of the voice disorder on their child (Zur et al., 2007). The pVHI consists of 23 items that parents complete using a five-point Likert scale (0: never, 1: almost never, 2: sometimes; 3: almost always; 4: always). Total pVHI scores range from 0 to 92 with a higher score corresponding with a greater impact.
  units on a scale | 20.73 (10.5) | 27.90 (11.1) | 23.50 (15.5) | 23.97 (12.2)
Consensus Auditory-Percpetual Evaluation of Voice - Overall Severity [Mean (Standard Deviation); unit: units on a scale] — The Consensus Auditory-Perceptual Evaluation of Voice is designed to describe the severity of dysphonia by rating six parameters (overall severity, roughness, breathiness, strain, pitch, and loudness) on a visual-analog scale from 0 to 100, where 0 is considered within normal limits. Overall Severity was selected as an outcome parameter.
  units on a scale | 22.67 (15.9) | 16.50 (5.1) | 32.50 (0.7) | 22.11 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Dysphonia Severity Index
Description: The dysphonia severity index (DSI) is a multiparametric score to quantify vocal capabilities. It is based on a weighted combination of 4 voice parameters: maximum phonation time (MPT, s), highest frequency (F-high, Hz), lowest intensity (I-low, dB) and jitter (%). The DSI is constructed as 0.13 MPT + 0.0053 F-high - 0.26 I-low - 1.18 jitter +12.4. The index ranges from -5 to +5. A score above +1.6 is considered normal. A higher score corresponds with better voice quality / vocal capacities.
Time Frame: pre: one day before therapy, day 0; post: immediately after last therapy session, day 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Experimental Group 1 - Straw Phonation | Experimental Group 2 - Resonant Voice Therapy | Control Group
Number analyzed (Participants) | 11 | 11 | 8
units on a scale | 1.8 [0.1 to 3.4] | 1.8 [0.1 to 3.4] | 0.0 [-1.9 to 1.9]
Statistical Analysis 1: Comparison: Experimental Group 1 - Straw Phonation vs Experimental Group 2 - Resonant Voice Therapy vs Control Group; Test type: Other; p = 0.024, Mixed Models Analysis — Linear Mixed Models: time-effect
Statistical Analysis 2: Comparison: Experimental Group 1 - Straw Phonation vs Experimental Group 2 - Resonant Voice Therapy vs Control Group; Test type: Other; p = 0.822, Mixed Models Analysis — Linear mixed models: group-effect
Statistical Analysis 3: Comparison: Experimental Group 1 - Straw Phonation vs Experimental Group 2 - Resonant Voice Therapy vs Control Group; Test type: Other; p = 0.290, Mixed Models Analysis — Linar mixed models: time*group-effect
Statistical Analysis 4: Comparison: Experimental Group 1 - Straw Phonation; Test type: Other; p = 0.035, Mixed Models Analysis — Linear mixed models: evolution pre-post; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [0.1 to 3.4]
Statistical Analysis 5: Comparison: Experimental Group 2 - Resonant Voice Therapy; Test type: Other; p = 0.038, Mixed Models Analysis — Linear mixed models: evolution pre-post; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [0.1 to 3.4]
Statistical Analysis 6: Comparison: Control Group; Test type: Other; p = 1.000, Mixed Models Analysis — Linear mixed models: evolution pre-post; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-1.9 to 1.9]

2. Primary Outcome: Change in Acoustic Voice Quality Index
Description: The acoustic voice quality index (AVQI) is a multiparametric score to quantify vocal quality. It is based on a weighted combination of 6 voice parameters: smoothed cepstral peak prominence (CPPS), harmonics-to-noise ratio (HNR), shimmer local (SL), shimmer local dB (SLdB), general slope of the spectrum (slope) and tilt of the regression line through the spectrum (tilt). The formula is constructed as 9.072 - 0.245 × CPPs - 0.161 × HNR - 0.470 × SL + 6.158 × SLdB - 0.071 × Slope - 0.170 × Tilt and ranges from 0 to 10. A lower score correlates with a better vocal quality.
Time Frame: pre: one day before therapy, day 0; post: immediately after last therapy session, day 4
Population: The audio samples of some participants were of insufficient quality to calculate the AVQI.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Experimental Group 1 - Straw Phonation | Experimental Group 2 - Resonant Voice Therapy | Control Group
Number analyzed (Participants) | 8 | 4 | 5
units on a scale | -0.1 [-0.6 to 0.4] | -0.4 [-1.1 to 0.3] | -0.3 [-0.9 to 0.3]
Statistical Analysis 1: Comparison: Experimental Group 1 - Straw Phonation vs Experimental Group 2 - Resonant Voice Therapy vs Control Group; Test type: Other; p = 0.107, Mixed Models Analysis — Linear mixed models: time-effect
Statistical Analysis 2: Comparison: Experimental Group 1 - Straw Phonation vs Experimental Group 2 - Resonant Voice Therapy vs Control Group; Test type: Other; p = 0.996, Mixed Models Analysis — Linear mixed models: group-effect
Statistical Analysis 3: Comparison: Experimental Group 1 - Straw Phonation vs Experimental Group 2 - Resonant Voice Therapy vs Control Group; Test type: Other; p = 0.639, Mixed Models Analysis — Linear mixed models: time*group-effect
Statistical Analysis 4: Comparison: Experimental Group 1 - Straw Phonation; Test type: Other; p = 0.731, Mixed Models Analysis — Linear mixed models: evolution pre-post; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.6 to 0.4]
Statistical Analysis 5: Comparison: Experimental Group 2 - Resonant Voice Therapy; Test type: Other; p = 0.217, Mixed Models Analysis — Linear mixed models: evolution pre-post; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.1 to 0.3]
Statistical Analysis 6: Comparison: Control Group; Test type: Other; p = 0.253, Mixed Models Analysis — Linear mixed models: evolution pre-post; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.9 to 0.3]

3. Primary Outcome: Change in Pediatric Voice Handicap Index (pVHI)
Description: The pediatric voice handicap index (pVHI) is a questionnaire to investigate children's voice-related quality of life, completed by the parents. The index ranges from 0 to 92. A higher score correlates with more psychosocial impact of the voice disorder.
Time Frame: pre: one day before therapy, day 0; post: immediately after last therapy session, day 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Experimental Group 1 - Straw Phonation | Experimental Group 2 - Resonant Voice Therapy | Control Group
Number analyzed (Participants) | 11 | 11 | 8
score on a scale | -3.3 [-7.2 to 0.7] | -3.9 [-8.3 to 0.4] | -1.7 [-6.7 to 3.2]
Statistical Analysis 1: Comparison: Experimental Group 1 - Straw Phonation vs Experimental Group 2 - Resonant Voice Therapy vs Control Group; Test type: Other; p = 0.024, Mixed Models Analysis — Linear mixed models: time-effect
Statistical Analysis 2: Comparison: Experimental Group 1 - Straw Phonation vs Experimental Group 2 - Resonant Voice Therapy vs Control Group; Test type: Other; p = 0.449, Mixed Models Analysis — Linear mixed models: group-effect
Statistical Analysis 3: Comparison: Experimental Group 1 - Straw Phonation vs Experimental Group 2 - Resonant Voice Therapy vs Control Group; Test type: Other; p = 0.786, Mixed Models Analysis — Linear mixed models: time*group-effect
Statistical Analysis 4: Comparison: Experimental Group 1 - Straw Phonation; Test type: Other; p = 0.099, Mixed Models Analysis — Linear mixed models: evolution pre-post; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-7.2 to 0.7]
Statistical Analysis 5: Comparison: Experimental Group 2 - Resonant Voice Therapy; Test type: Other; p = 0.074, Mixed Models Analysis — Linear mixed models: evolution pre-post; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-8.3 to 0.4]
Statistical Analysis 6: Comparison: Control Group; Test type: Other; p = 0.472, Mixed Models Analysis — Linear mixed models: evolution pre-post; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-6.7 to 3.2]

4. Primary Outcome: Change in Overall Severity From Consensus Auditory-Perceptual Evaluation of Voice
Description: This tool is designed to describe the severity of dysphonia by rating six parameters (overall severity, roughness, breathiness, strain, pitch, and loudness) on a visual-analog scale from 0 to 100, where 0 is considered within normal limits. A higher score corresponds with worse voice quality.
Time Frame: pre: one day before therapy, day 0; post: immediately after last therapy session, day 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Experimental Group 1 - Straw Phonation | Experimental Group 2 - Resonant Voice Therapy | Control Group
Number analyzed (Participants) | 11 | 11 | 8
score on a scale | -6.5 [-12.2 to -0.9] | -0.7 [-6.4 to 4.9] | -1.0 [-7.7 to 5.7]
Statistical Analysis 1: Comparison: Experimental Group 1 - Straw Phonation vs Experimental Group 2 - Resonant Voice Therapy vs Control Group; Test type: Other; p = 0.115, Mixed Models Analysis — Linear mixed models: time-effect
Statistical Analysis 2: Comparison: Experimental Group 1 - Straw Phonation vs Experimental Group 2 - Resonant Voice Therapy vs Control Group; Test type: Other; p = 0.516, Mixed Models Analysis — Linear mixed models: group-effect
Statistical Analysis 3: Comparison: Experimental Group 1 - Straw Phonation vs Experimental Group 2 - Resonant Voice Therapy vs Control Group; Test type: Other; p = 0.276, Mixed Models Analysis — Linear mixed models: time*group-effect
Statistical Analysis 4: Comparison: Experimental Group 1 - Straw Phonation; Test type: Other; p = 0.025, Mixed Models Analysis — Linear mixed models: evolution pre-post; Mean Difference (Final Values) = -6.5, 95% CI 2-sided [-12.2 to -0.9]
Statistical Analysis 5: Comparison: Experimental Group 2 - Resonant Voice Therapy; Test type: Other; p = 0.794, Mixed Models Analysis — Linear mixed models: evolution pre-post; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-6.4 to 4.9]
Statistical Analysis 6: Comparison: Control Group; Test type: Other; p = 0.760, Mixed Models Analysis — Linear mixed models: evolution pre-post; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-7.7 to 5.7]

ADVERSE EVENTS:
Time Frame: 3 months after completion of the voice therapy program
Description: Definitions did not differ from the clinicaltrials.gov definitions.
Arm/Group | Experimental Group 1 - Straw Phonation | Experimental Group 2 - Resonant Voice Therapy | Control Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/8

LIMITATIONS AND CAVEATS:
It was not possible to analyze the long-term results due to high drop-out.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT05878197/Prot_SAP_000.pdf